CLINICAL TRIAL: NCT02754375
Title: Cerebral Functional Modifications After Low Frequency Repetitive Transcranial Magnetic Stimulation in Refractory Depression. Assessment With 18F-FDG-PET Imaging.
Brief Title: SMTr-METAB : FDG-PET Assessment of Cerebral Metabolism in Resistant Depression Treated With rTMS
Acronym: SMTr-METAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-PP-02
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Depression
Keywords: biological markers; rTMS
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient (Experimental): Patient with resistant depression treated with rTMS
  Interventions: Procedure: rTMS

INTERVENTIONS:
Procedure: rTMS

SUMMARY:
Biological markers of depressive states have been studied, but their usefulness to predict the therapeutic response is unknown. This issue is major in all depressive states which have not remitted after several lines of treatment. rTMS (repetitive transcranial magnetic stimulation) is a non-pharmacological alternative in the treatment of depression, but its effects on cerebral functioning are not known in episodes which have resist to conventional treatments. The investigators will include 50 depressive patients who have failed to respond to two successive antidepressant medication, and propose them a treatment with low frequency rTMS during 3 to 6 weeks. Cerebral functional imaging with 18FDG-PET (positon emission tomography) with be assessed at the beginning and at the end of rTMS acute treatment, in order to measure induced metabolic changes and their correlation with clinical states. Patients who have responded to rTMS acute treatment may continue this therapeutic for six months, and the investigators will assess if efficacy maintenance is related with cerebral metabolic variations

DETAILED DESCRIPTION:
In France, lifetime prevalence of depression is 21 %, with major consequences: handicap, loss of productivity, reduction in quality of life, increased mortality. The efficient and long-lasting care of depression is consequently a priority of public health.

Despite well-conducted conventional therapeutic strategies, it is estimated that about 30 % of the depressed patients do not respond at all to an antidepressant, that 30 % will present a partial response, and that 40 % only patients will have a complete remission.

Non-pharmacological alternative treatments have been promoted, particularly with repetitive transcranial magnetic stimulation (rTMS). A recent meta-analysis with 29 randomized controlled trials versus placebo reports a 29.3 % response rate and a 18.6 % remission rate after active stimulation vs respectively, 10.4 % and 5 % after placebo stimulation.

However, predictive biomarkers of response are unknown, and cerebral metabolism may be a good candidate. It is admitted that the depressive state is correlated with specific modifications of glucose metabolism in circuits which are involved in the neurobiology of depression. The amplitude of these changes may correlate with clinical severity or may differ with treatment type, and cerebral metabolic changes might be an additional guide to treatment. Finally, the therapeutic effect might normalize cerebral functional activity and this might be an early correlate of clinical response. However the studies using functional imaging in a therapeutic approach or in the understanding of the physiopathology of the depression are not usable in a clinical practice of routine.

The investigators suggest using a well-known analysis software (Scenium software, Siemens GmbH) who allows an automated analysis by the distribution of the cerebral metabolism by means of the F18-FDG TEP-TDM and a quantitative measure, expressed in regional consumption of glucose expressed by g / 100 g / min for every 18F-FDG TEP-TDM and for every region of interest. Image registering by the camera, remote of the injection of the tracer, lasts less than 10 minutes.The software also allows to compare the data acquired for a patient with a standardized database.

The investigators will perform a opened study in two centers (Monaco Hospital/Nice CHU) on 50 depressed patients aged from 40 to 65 years old, not having answered 2 lines of well led antidepressants. Low-frequency rTMS will be proposed in acute cure (3 in 6 weeks) in monotherapy followed by 6 months of rTMS for patients who have responded to acute treatment phase.

Cerebral metabolic modifications (location and intensity) will be calculated after two PET-TDM in every patient, realized before and after the acute treatment by rTMS. We shall use the SCENIUM software which allows to compare each patient's data with a standardized database.

At the end of the acute period of treatment, it will be proposed to patients who have responded to pursue rTMS treatment in a consolidation phase for 6 months. All patients will be longitudinally assessed during this consolidation period. One objective is to assess if initial TEP-TDM data and/or the amplitude of the induced metabolic variation is associated with the stability of the clinical answer in respondent patients

ELIGIBILITY:
Inclusion Criteria:

* Subject from 40 to 65 years old
* Characterized current depressive Episode, unipolar, without psychotic characteristic (according to DSM IV-TR)
* Presenting to the inclusion a score upper or equal to 20 on the scale HDRS-17
* Absence of answer or partial clinical answer to more than two antidepressant treatments of different therapeutic classes to effective posology on a duration of at least 6 weeks
* Patient affiliated to French social security
* Patient must give a written, signed and dated informed consent before any study related activity is performed. Where relevant, a legal representative will also sign the informed study consent according to local laws and regulations

Exclusion Criteria:

* Failure in a previous low-frequency rTMS cure (at least 15 sessions)
* Failure in a cure of bilateral ECT (at least 8 sessions) or unilateral (at least 10 sessions)
* Mental disorder owed to a general medical affection ( DSM-IV)
* Presence of a neurodegenerative pathology in the inclusion estimated on the clinical examination, the intellectual MRI, the TEP / TDM at the 18F-FDG and the neuropsychological profile in the inclusion
* Severe or not stabilized somatic Disease
* chronic depression evolving for more than 3 years
* Not answer in more of therapeutic antidepressive five well (documented) conducts
* Presence of contraindication the SMTr, of which epileptic disease
* Schizophrenic Disorder
* Addicting Disorder with current dependence (alcohol, cannabis, benzodiazepin)
* Bipolar disorder (I, II)
* Disorder of personality to cluster A and B co-morbid
* Pregnant Woman (dosage of urinary Beta-HCG)
* Vulnerable Person: major under guardianship or guardianship, minor
* Mental Deficiency of the subject making its participation on approval impossible
* Participation in another clinical trial

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Variation of the regional cerebral glucose consumption between the two PET-TDM | at week 6
  Variation of the regional cerebral glucose consumption between the two PET-TDM (realized at inclusion and at Week 6)

SECONDARY OUTCOMES:
Comparison of local glucose use between responder and non-responder patients | at week 6

CONTACTS AND LOCATIONS:
Locations (2):
- CHU de Nice, Nice, France
- Hôpital Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No